CLINICAL TRIAL: NCT00500318
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 6-Week Clinical Study to Assess the Effect of Inhaled Aclidinium Bromide (LAS34273) 200 ug on Exercise Endurance and Lung Hyperinflation in Patients With Moderate to Severe COPD
Brief Title: A Study of Exercise Endurance and Lung Hyperinflation in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAS-MD-CL26
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Bronchitis, Chronic; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Bronchiolitis Obliterans Syndrome; Emphysema | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Aclidinium (Experimental)
  Interventions: Drug: Aclidinium Bromide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium Bromide — Aclidinium Bromide, 200μg. Once daily oral inhalation.
  Arms: Aclidinium
Drug: Placebo — Dose matched placebo, once daily oral inhalation.
  Arms: Placebo

SUMMARY:
This study evaluated the effect of inhaled aclidinium bromide on exercise endurance and in reducing resting and dynamic lung hyperinflation in patients with moderate to severe COPD. It was 9 weeks in duration, consisting of; a 2-week run-in period, 6 weeks of double-blind treatment, and a 1-week follow-up phone call. All patients meeting the eligibility criteria were randomized to one of two treatment groups: aclidinium bromide or placebo.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of stable moderate to severe COPD (GOLD 2006); post-levalbuterol FEV1 >=30% and < 80% predicted and FEV1/FVC<70% predicted
* Current or former cigarette smoker
* Functional Residual Capacity (FRC) measured by body plethysmography >= 120% of predicted value
* Baseline Dyspnea Index (BDI) focal score ≤ 7 at Visit 4

Exclusion Criteria:

* History of presence of asthma, allergic rhinitis, or atopy
* Hospitalization for acute COPD exacerbation in the 3 months prior to study entry
* Respiratory tract infection (including the upper respiratory tract) or COPD exacerbation in the 6 weeks prior to study entry
* Clinically significant respiratory conditions other than COPD
* Chronic use of oxygen therapy >= 15 hours a day

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (52):
- United States (42):
  - Forest Investigative Site 2088, Jasper, Alabama
  - Forest Investigative Site 0909, Phoenix, Arizona
  - Forest Investigative Site 0957, Long Beach, California
  - Forest Investigative Site 0973, Los Angeles, California
  - Forest Investigative Site 0887, Los Angeles, California
  - Forest Investigative Site 0988, Sacramento, California
  - Forest Investigative Site 0885, Torrance, California
  - Forest Investigative Site 2663, Clearwater, Florida
  - Forest Investigative Site 1030, Jacksonville, Florida
  - Forest Investigative Site 0974, Pensacola, Florida
  - Forest Investigative Site 0980, Atlanta, Georgia
  - Forest Investigative Site 0991, Atlanta, Georgia
  - Forest Investigative Site 0987, Austell, Georgia
  - Forest Investigative Site 2008, Marietta, Georgia
  - Forest Investigative Site 0984, Iowa City, Iowa
  - Forest Investigative Site 1080, Topeka, Kansas
  - Forest Investigative Site 0898, Baltimore, Maryland
  - Forest Investigative Site 0886, Boston, Massachusetts
  - Forest Investigative Site 1029, North Dartmouth, Massachusetts
  - Forest Investigative Site 0889, Livonia, Michigan
  - Forest Investigative Site 2079, Saint Charles, Missouri
  - Forest Investigative Site 2071, Omaha, Nebraska
  - Forest Investigative Site 0972, Brooklyn, New York
  - Forest Investigative Site 0971, Great Neck, New York
  - Forest Investigative Site 1114, New York, New York
  - Forest Investigative Site 2665, New York, New York
  - Forest Investigative Site 2081, Charlotte, North Carolina
  - Forest Investigative Site 0688, Charlotte, North Carolina
  - Forest Investigative Site 0981, Toledo, Ohio
  - Forest Investigative Site 1057, Hershey, Pennsylvania
  - Forest Investigative Site 0888, Philadelphia, Pennsylvania
  - Forest Investigative Site 0983, Scranton, Pennsylvania
  - Forest Investigative Site 2072, Charleston, South Carolina
  - Forest Investigative Site 1107, Columbia, South Carolina
  - Forest Investigative Site 0979, Columbia, South Carolina
  - Forest Investigative Site 1078, Greenville, South Carolina
  - Forest Investigative Site 0900, Spartanburg, South Carolina
  - Forest Investigative Site 0962, Nashville, Tennessee
  - Forest Investigative Site 1082, Dallas, Texas
  - Forest Investigative Site 2058, Dallas, Texas
  - Forest Investigative Site 0890, Houston, Texas
  - Forest Investigative Site 0977, Midvale, Utah
- Canada (10):
  - Forest Investigative Site 0968, Edmonton, Alberta
  - Forest Investigative Site 0960, Kelowna, British Columbia
  - Forest Investigative Site 0905, Vancouver, British Columbia
  - Forest Investigative Site 0976, Winnipeg, Manitoba
  - Forest Investigative Site 0891, Hamilton, Ontario
  - Forest Investigative Site 2204, Ottawa, Ontario
  - Forest Investigative Site 0969, Windsor, Ontario
  - Forest Investigative Site 2205, Montreal, Quebec
  - Forest Investigative Site 0893, Ste-Foy, Quebec
  - Forest Investigative Site 0943, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Maltais F, Celli B, Casaburi R, Porszasz J, Jarreta D, Seoane B, Caracta C. Aclidinium bromide improves exercise endurance and lung hyperinflation in patients with moderate to severe COPD. Respir Med. 2011 Apr;105(4):580-7. doi: 10.1016/j.rmed.2010.11.019. Epub 2010 Dec 22. PMID 21183326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from July to October of 2007 at 52 study sites (42 sites in the United States and 10 additional sites in Canada)
Pre-assignment Details: All demographic and baseline characteristics were analyzed descriptively just for the Safety population.
Groups:
- Aclidinium: Aclidinium bromide, 200 micrograms, oral inhalation once per day.
- Placebo: Dose-matched placebo, oral inhalation, once per day.
Period: Overall Study
Arm/Group | Aclidinium | Placebo
Started | 86 | 95
Completed | 81 | 78
Not Completed | 5 | 17
Not completed — Adverse Event | 3 | 8
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 0 | 3
Not completed — Other Reason | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium | Placebo | Total
Number analyzed (Participants) | 86 | 95 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.5) | 65.6 (7.8) | 64.8 (8.6)
Gender [Count of Participants; unit: Participants]
  Female | 34 | 42 | 76
  Male | 52 | 53 | 105
Region of Enrollment [Number; unit: participants]
  United States | 64 | 75 | 139
  Canada | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Exercise Endurance Time (ET)
Description: Exercise endurance time is defined as the time from the increase in work rate at 75% Wmax (watts) to the point of symptom limitation. The Wmax is defined as the highest work rate the patients were able to maintain for at least 30 seconds.
Time Frame: From baseline Week 0 (Visit 4) to Week 6 (Visit 6)
Population: Missing data for patients who withdrew due to COPD exacerbations was imputed using the Worst Observation Carried Forward (WOCF) of all Endurance time (ET), while ETs that were missing for other reasons were imputed using the Last Observation Carried Forward (LOCF) method based on the last visit available.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 86 | 94
Seconds | 129.45 (31.19) | 13.01 (30.97)
Statistical Analysis 1: Comparison: Aclidinium vs Placebo; Test type: Superiority or Other; p = 0.0042, ANCOVA; Least Square Mean = 116.44, 95% CI 2-sided [37.280 to 195.610], Standard Error of Mean 40.113

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in trough Forced Expiratory Volume in 1 second. FEV1 was assessed at the end of the daily dosing interval (Trough).
Time Frame: Change from baseline (Visit 4) at Week 6 (Visit 6)
Population: The Intent-to-Treat (ITT) population consisted of all patients in the Safety Population who had at least a baseline and one post-baseline assessment of the primary efficacy parameter. Missing values due to a premature discontinuation or patients who missed specific trial visits were imputed by Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 86 | 92
L | 0.090 (0.018) | -0.010 (0.018)

3. Secondary Outcome: Trough Inspiratory Capacity (IC)
Description: Change in trough Inspiratory Capacity. Inspiratory Capacity was measured as part of the spirometry procedures performed at each visit. IC was assessed at the end of the daily dosing interval (Trough).
Time Frame: Change from baseline Week 0 (Visit 4) to Week 6 (Visit 6)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 83 | 90
L | 0.083 (0.032) | -0.019 (0.032)

4. Secondary Outcome: Functional Residual Capacity (FRC)
Description: Change in trough Functional Residual Capacity. FRC was assessed at the end of the daily dosing interval (Trough).
Time Frame: Change from baseline Week 0 (Visit 4) to Week 6 (Visit 6)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 81 | 78
L | -0.138 (0.061) | -0.076 (0.064)

5. Secondary Outcome: Inspiratory Capacity (IC)/Total Lung Capacity (TLC) Ratio
Description: Ratio of trough Inspiratory Capacity verses Total Lung Capacity.
Time Frame: Change from baseline Week 0 (Visit 4) to Week 6 (Visit 6)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Aclidinium | Placebo
Number analyzed (Participants) | 78 | 75
ratio | 0.014 (0.006) | -0.003 (0.006)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from July of 2007 to December of 2008 at 52 study sites (42 sites in the United States and 10 additional sites in Canada)
Arm/Group | Aclidinium | Placebo
Serious Adverse Events (participants affected / at risk) | 2/86 | 3/95
Other Adverse Events (participants affected / at risk) | 16/86 | 18/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium (N=86) | Placebo (N=95)
Ileitis (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium (N=86) | Placebo (N=95)
Headache (Nervous system disorders) | 5 | 7
Chronic Obstructive Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of the Sponsor. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and the Sponsor.